CLINICAL TRIAL: NCT01705925
Title: Multicenter Evaluation of Children and Young Adults With Genotype Positive Long QT Syndrome
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: PDX-002-11
Record Dates: First submitted 2012-10-04; First posted 2012-10-12 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Long QT Syndrome
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to provide comprehensive follow-up in patients with Long QT Syndrome (LQTS) and gain additional information regarding genotype-phenotype correlation and effective management and treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Children and/or young adults diagnosed with heterogeneous repolarization disorder who have genotype positive Long QT, or
* Newly diagnosed mutation positive patients with a confirmed test

Exclusion Criteria:

* Children who are phenotypically positive with no molecular testing
* Children that are phenotypically positive but genotype negative

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and Young Adults with Genotype Positive Long QT Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Adverse Cardiac Events on patients with genotype positive LQT1 who have a normal EKG and absence of symptoms, but a molecular confirmation of LQT1. | Enrollment is expected to take approximately 5 years. The patients will be followed until they are no longer cared for by a pediatric cardiology facility (typically post-college) or approximately 21 years of age.

SECONDARY OUTCOMES:
Adverse Cardiac Events on patients with both phenotype and genotype positive. | Enrollment is expected to take approximately 5 years. The patients will be followed until they are no longer cared for by a pediatric cardiology facility (typically post-college) or approximately 21 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cohen, M.D., Principal Investigator — Pediatrix; Arnold Fenrich, MD, Principal Investigator — Pediatrix; Reese Clark, MD, Study Director — Pediatrix
Locations (1):
- Children's Cardiology Associates, Austin, Texas, United States